CLINICAL TRIAL: NCT02166983
Title: Cognitive Enhancement Program
Brief Title: Cognitive Enhancement Program in Improving Cognitive Function in Breast Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left Stanford
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BRS0037; NCI-2013-02353 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRS0037 (Other: Stanford University Hospitals and Clinics); P30CA124435 (NIH)
Record Dates: First submitted 2013-12-16; First posted 2014-06-18 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer; Cancer Survivor; Cognitive/Functional Effects
MeSH Terms: conditions — Breast Neoplasms | interventions — Mind-Body Therapies

ARMS (3):
- Arm IA (Lumosity, relaxation, compensatory strategies) (Experimental): Participants complete Lumosity cognitive exercises. Lumosity cognitive exercises are online video game-based activities that are designed to practice various cognitive skills including processing speed, attention, memory and executive function. Participants complete cognitive exercises at least 20 minutes a day, 5 days a week for 6 weeks. Participants also complete relaxation exercises (guided imagery, progressive muscle relaxation, and/or autogenics) at least 10 minutes a day for 6 weeks and compensatory strategies (the use of external devices such as a notebook, day planner, or smartphone for cuing, reminding, and organizing; the use of memory strategies such as repetition, paraphrasing, and active listening; and the use of executive strategies such as self-talk for planning and attention orientation) as much as possible.
  Interventions: Other: computer-assisted cognitive training; Procedure: mind-body intervention procedure; Other: memory intervention; Other: questionnaire administration
- Arm IB (Active Journaling, relaxation, compensatory strategy) (Experimental): Participants complete Active Journal cognitive exercises. Active Journaling requires participants to keep a written diary or journal where she discusses what her thoughts and feelings about various events with a focus on describing the meaning of the activities and experiences, particularly new things that were learned. Active Journaling is a method of practicing various cognitive skills including communication, organization, memory and executive function. Participants complete cognitive exercises at least 20 minutes a day, 5 days a week for 6 weeks. Participants also complete relaxation exercises and compensatory strategies as in Arm IA.
  Interventions: Other: cognitive intervention; Procedure: mind-body intervention procedure; Other: memory intervention; Other: questionnaire administration
- Arm II (Lumosity only) (Experimental): Participants complete Lumosity exercises as in Arm IA.
  Interventions: Other: computer-assisted cognitive training; Other: questionnaire administration

INTERVENTIONS:
Other: computer-assisted cognitive training — Complete Lumosity cognitive exercises
  Arms: Arm IA (Lumosity, relaxation, compensatory strategies); Arm II (Lumosity only)
Other: cognitive intervention — Complete Active Journaling cognitive exercises
  Arms: Arm IB (Active Journaling, relaxation, compensatory strategy)
Procedure: mind-body intervention procedure — Complete relaxation exercises
  Other Names: mind-body interventions
  Arms: Arm IA (Lumosity, relaxation, compensatory strategies); Arm IB (Active Journaling, relaxation, compensatory strategy)
Other: memory intervention — Complete compensatory strategies
  Arms: Arm IA (Lumosity, relaxation, compensatory strategies); Arm IB (Active Journaling, relaxation, compensatory strategy)
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies cognitive enhancement program in improving cognitive function in breast cancer survivors. A cognitive enhancement program may help improve cognitive function in breast cancer survivors and may help doctors plan better treatment for cognitive decline.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To improve cognition of women who have had breast cancer and exhibit cognitive decline through a cognitive enhancement program.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I (Cognitive Enhancement Program): Participants are randomized to 1 of 2 arms.

ARM IA (Lumosity): Participants complete Lumosity cognitive exercises. Lumosity cognitive exercises are online video game-based activities that are designed to practice various cognitive skills including processing speed, attention, memory and executive function. Participants complete cognitive exercises at least 20 minutes a day, 5 days a week for 6 weeks. Participants also complete relaxation exercises (guided imagery, progressive muscle relaxation, and/or autogenics) at least 10 minutes a day for 6 weeks and compensatory strategies (the use of external devices such as a notebook, day planner, or smartphone for cuing, reminding, and organizing; the use of memory strategies such as repetition, paraphrasing, and active listening; and the use of executive strategies such as self-talk for planning and attention orientation) as much as possible.

ARM IB (Active Journaling): Participants complete Active Journal cognitive exercises. Active Journaling requires participants to keep a written diary or journal where she discusses what her thoughts and feelings about various events with a focus on describing the meaning of the activities and experiences, particularly new things that were learned. Active Journaling is a method of practicing various cognitive skills including communication, organization, memory and executive function. Participants complete cognitive exercises at least 20 minutes a day, 5 days a week for 6 weeks. Participants also complete relaxation exercises and compensatory strategies as in Arm IA.

ARM II (Lumosity only): Participants complete Lumosity cognitive exercises as in Arm IA.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of breast cancer
* Received chemotherapy treatment for breast cancer diagnosis
* Chemotherapy-free for at least one year

Exclusion Criteria:

* History of learning disability, head trauma, neurologic disorder or significant psychiatric condition
* Significant medical condition (e.g. diabetes) unrelated to cancer diagnosis
* Magnetic resonance imaging (MRI) contraindications (e.g. metallic biomedical implants)
* Pregnancy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Standardized Executive Function Test Composite Score | Baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shelli Kesler, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States